CLINICAL TRIAL: NCT03113097
Title: Does Transfer of Poor-quality Embryos With Good-quality Embryos Improve Pregnancy Outcome in Women Undergoing IVF/ICSI?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Collaborators: Dar El Teb Institute (Other)
Responsible Party: Principal Investigator, Mohammed Faris, Dr Mohammed Faris, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DAT-055
Record Dates: First submitted 2017-04-10; First posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Embryo Transfer

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Good-quality embryo transfer (Active Comparator): Women who had only good-quality embryo transfer
  Interventions: Other: Embryo transfer
- good- and poor-quality embryo transfer (Active Comparator): Women who had both good- and poor-quality embryo transfer
  Interventions: Other: Embryo transfer

INTERVENTIONS:
Other: Embryo transfer — Transfer of different qualities of embryos at blastocyst stage

SUMMARY:
Women planned to undergo blastocyst-stage embryo transfer after IVF/ICSI were randomized into 2 groups:

* group I: women who had only good-quality embryo transfer.
* group II: women who had both good-quality and poor-quality embryo transfer.

primary outcome was ongoing clinical pregnancy rate

ELIGIBILITY:
Inclusion Criteria:

* women undergoing primary IVF/ICSI cycles for tubal factor/unexplained infertility and had blastocyst-stage ET

Exclusion Criteria:

* cleavage-stage ET.
* women who had no good-quality embryos to transfer
* women who had known poor endometrial receptivity

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 627 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Ongoing clinical pregnancy rate | 12 weeks
  viable intrauterine pregnancy ongoing beyond 12 weeks of gestation

SECONDARY OUTCOMES:
Biochemical pregnancy rate | 2 weeks after ET
  positive serum hCG
Clinical pregnancy rate | 4 weeks after ET
  sonographic detection of viable intrauterine gestational sac
Multiple pregnancy rate | 4-6 weeks after ET
  No. of intrauterine gestational sacs
Ectopic pregnancy rate | 6 weeks after ET
  Extrauterine pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Faris, MD, Principal Investigator — Dar El Teb IVF and Infertility Center